CLINICAL TRIAL: NCT05291169
Title: A Randomized, Multicenter, Open Label Study Comparing Omeza Combination Therapy With Standard of Care to Standard of Care Alone for Chronic Venous Leg Ulcers
Brief Title: Omeza Combination Therapy With Standard of Care to Standard of Care Alone for Chronic Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OM-CTP-001.1
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized to Omeza Combination therapy and SOC Vs SOC alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OCM™ plus Standard of Care (Experimental): Omeza® OCM™ is an FDA cleared 510(K) medical combination drug/device which is applied directly to the wound bed. Treatment, followed by compression management, is applied on a weekly basis.
  Interventions: Device: Omeza® OCM™
- Standard of Care (No Intervention): Cleaning and debridement of the ulcers with compression management on a weekly basis.

INTERVENTIONS:
Device: Omeza® OCM™ — Omeza® OCM™ is a wound care matrix comprised of coldwater fish peptides (device) and cod liver oil (drug).
  OCM™is supplied in a sterile single use vial.
  Other Names: Omeza® Complete Matrix; Multimodal Wound Matrix
  Arms: OCM™ plus Standard of Care

SUMMARY:
A Randomized, Multicenter, Open Label Study Comparing Omeza Combination Therapy with Standard of Care to Standard of Care alone for Chronic Venous Leg Ulcers over the course of 4 weeks

DETAILED DESCRIPTION:
The study will have three phases: Screening, Treatment and Healing Confirmation.

The Screening Phase (1 -14 days) is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study and consists of a series of screening assessments designed to determine eligibility.

At or up to 14 days before the first Screening Phase Visit (S1), written informed consent from the subject will be obtained by the Investigator or suitably qualified designee before the performance of any other protocol-specific procedure.At the first Screening Phase Visit (S1), the Investigator will select the study (target) ulcer. Each subject will have only one VLU selected as the study (target) ulcer. In the situation where a subject has more than one VLU at the S1 visit, the Investigator will select the largest VLU that meets the eligibility criteria of the protocol as the study (target) ulcer.

Subjects whose target ulcer has been treated with compression therapy for the previous two weeks are eligible to enter the treatment phase once all of the inclusion and exclusion criteria are met. Note: if the target ulcer has not received any high-strength compression, the subject must be placed into compression for a minimum of 14 days prior to enrollment (run-in phase).

The Treatment Phase (TV1 to TV4) begins with a series of assessments designed to confirm the subject's continued eligibility. Subjects whose ulcers continue to meet eligibility criteria will then be randomized to one of two groups: (1) Omeza Combination Therapy (a lidocaine based periulcer preparation, a collagen-based topical treatment, and a periwound protectant) plus Standard of Care; or (2) Standard of Care (multiple layered compression therapy) alone.

At the conclusion of the 4-week treatment visits, enrolled Subjects will have the option to continue receiving Omeza Combination Therapy and Standard of Care protocol up to an additional 8 weeks.

Assessments will be taken and further therapy for the Subject will be at the PI's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old and female subjects are not pregnant
2. Study ulcer has been present for at least 1 month and less than or equal to 12 months as of the date the subject signs consent for study
3. Study ulcer size is a minimum of 4.0 cm2 and a maximum of 100.0 cm2
4. The ulcer must be between the knee and ankle, at or above the malleolus, and full thickness without exposed muscle, tendon, or bone
5. Known HbA1c of < 10% within 3 months
6. Study ulcer may have characteristics that include yellow/white slough with or without fibrous/scar tissue and/or non-viable tissue, but not mandatory
7. If more than one ulcer is present on the same leg, they must be greater than 2 cm apart and only the larger ulcer will be included in the study
8. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within (1 or 2) months of the first screening visit are acceptable:

   1. ABI between 0.8 and ≤ 1.3
   2. TBI ≥ 0.6
   3. TCOM ≥ 40 mmHg
   4. PVR: biphasic or triphasic waveforms
9. Subject understands and is willing to participate in the clinical study including compression for minimum 14 days (compression dressing changed once weekly) prior to study start (see page 23), participate in the informed consent process, and can comply with weekly visits and the Version 1 Confidential Page 8 of 51 follow-up regimen
10. Willing and able to comply with study procedures, including study visits and study dressing regimens (or have family member/friend willing and able), including ability of the subject to tolerate limb compression bandage
11. Subject has read and signed the IRB-approved Informed Consent Form before screening procedures are undertakenExclusion Criteria:

Exclusion

1. Study ulcer deemed by the Investigator to be caused by a medical condition other than venous insufficiency.
2. Study ulcer exhibits clinical signs and symptoms of infection, as evidenced by tissue necrosis, redness, pain, and/or purulent drainage and/or receiving systemic antibiotics for the treatment of such
3. Study ulcer is treated with a topical antibiotic during the screening phase.
4. Study ulcer requires enzymatic debridement during the study.
5. Study ulcer has undergone 12 or more months of continuous high-strength compression therapy over its duration.
6. Study ulcer is less than 4.0 cm2 or greater than 100.0 cm2 (Determined by MolecuLight Imaging Device).
7. Study ulcer extends more than 50% below the malleolus.
8. Study ulcer has been treated with tissue engineered material (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g., Oasis, PuraPly AM or Matristem) within the last 30 days.
9. Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
10. Study ulcer decreases in area by 30% or more during the 14 days screening period.
11. Subjects who are unable to understand the aims and objectives of the trial or have a known history of poor adherence with medical treatment.
12. Presence of any condition(s) that seriously compromises the subject's ability to complete this study.
13. Subjects with a BMI>65
14. Subject is an active smoker
15. Subject has any history of fish allergy or a known sensitivity to any of the SoC materials which come into contact with the skin
16. Ankle-Branchial Index (ABI) less than 0.80 or greater than 1.3
17. Presence of any monophasic waveforms on segmental Arterial Doppler/Pulse Volume Recording
18. Subject is on Dialysis
19. Any active cancer other than a nonmelanoma skin cancer; any previous cancer must be in remission for at least 1 year: bone cancer of metastatic disease of the affected limb, or has had chemotherapy within the last 12 months
20. Suspicion of malignancy within VLU. Any wound that has been present for > 6 months and hasn't previously been biopsied, a biopsy must be performed. Also, if a clinical suspicion of malignancy exists in the opinion of the Investigator, a biopsy should be performed regardless of duration of wound.
21. Life expectancy < 6 months
22. Subject has received within 28 days of screening a treatment which is known to interfere with or affect the rate and quality of wound healing (e.g., thrombolysis, systemic steroids, immunosuppressive therapy, autoimmune disease therapy, dialysis, radiation therapy,chemotherapy, revascularization surgery) to the leg or who may receive such medications during the screening period or who has anticipated to require such medications during the course of the study.
23. History of immunodeficiency or any illness or condition that could interfere with wound healing e.g., lymphedema, end-stage renal disease, severe malnutrition, liver disease, aplastic anemia. Raynaud's Syndrome, connective tissue disorder, acquired immune deficiency syndrome, HIV positive, or sickle cell anemia
24. Untreated osteomyelitis
25. Hepatitis
26. Acute deep venous thrombosis
27. Allergy to lidocaine and/or epinephrine
28. Subject's inability to successfully tolerate compression therapy that is changed weekly
29. All females of childbearing potential who are not using a highly effective method of birth control (failure rate less than 1% per year), such as implants, injectables, combined oral contraceptives, some IUDs, practice sexual abstinence or have a vasectomized partner.
30. The following are prohibited within 30 days prior to randomized treatment and throughout the study

1. Heat lamps 2. UV lights 3. Whirlpool baths 4. Hyperbaric oxygen 5. Jet water streams (other than gentle saline irrigation)

*Note: an ulcer that is deemed infected at S1 or TV1 might be eligible for re-screening once the infection is resolved, at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile of the Omeza Combination Therapy for chronic venous leg ulcers | 12 weeks
  To evaluate the safety profile of the Omeza Combination Therapy for chronic venous leg ulcers through SAE/AE reporting
To evaluate the impact on chronicity of wound healing by Omeza Combination Therapy and Standard of Care (multilayer compression) at week 4 compared to Standard of Care | 4 weeks
  To evaluate the impact on chronicity of wound healing by Omeza Combination Therapy and Standard of Care (multilayer compression) at week 4 compared to Standard of Care by Wound measurements using the MolecuLight Imaging Device
To evaluate change in ulcer size at week 4 (percent area reduction) compared to baseline | 4 weeks
  To evaluate change in ulcer size at week 4 (percent area reduction) compared to baseline based on wounds measurements using the MolecuLight Imaging Device

SECONDARY OUTCOMES:
Change in the subjects' Quality of Life (QoL) a. week to week using a numerical scale b. reported pain perception c. assessment of drainage d. enhanced activities in daily living | 12 weeks
  Change in the subjects' Quality of Life (QoL) using the PEG scale which is a validated pain scoring system. It consists of three 1-10 rating scales: numerical, enjoyment of life and general activity. The subject indicates a numerical value that best represents the pain intensity at ulcer site on a scale of 0 to 10 anchored by word descriptors at each end, as "no pain" on the left side and "Pain as bad as you can imagine" on the right side of the number line.

OTHER OUTCOMES:
Change in bacterial fluorescence using the MolecuLight device at baseline and weekly. | 12 weeks
  Change in bacterial fluorescence using the MolecuLight device at baseline and weekly at their weekly treatment visits

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, FACS, Study Chair — SerenaGroup, Inc.; Desmond Bell, DPM, Study Director — Omeza, LLC
Locations (7):
- United States (7):
  - New Hope Podiatry, Los Angeles, California
  - Royal Research, Corp, Hollywood, Florida
  - Three Rivers Wound and Hyperbaric Center, North Port, Florida
  - Wound Care of Tulsa, Tulsa, Oklahoma
  - The Foot and Ankle Wellness Center of Western Pennsylvania, Ford City, Pennsylvania
  - ACMH Wound Clinic, Kittanning, Pennsylvania
  - Serena Group, Monroeville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No